CLINICAL TRIAL: NCT04508036
Title: The Relationship of Ductus Arteriosus Closure and D-Dimer and Fibrinogen Levels in Premature Babies
Brief Title: Ductus Arteriosus Closure and D-Dimer and Fibrinogen Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, Associate Professor of Neonatology, Hacettepe University
Other Study IDs: KA-19033
Record Dates: First submitted 2020-08-01; First posted 2020-08-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Ductus Arteriosus, Patent
Keywords: Premature Newborn; Ductus Arteriosus; D-Dimer; Fibrinogen
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Premature newborns born before 32nd gestational week and weighing less than 1500 grams.
  Interventions: Diagnostic Test: Withdrawal of blood samples for D-Dimer; Diagnostic Test: Withdrawal of blood samples for Fibrinogen; Diagnostic Test: Echocardiographic Examination

INTERVENTIONS:
Diagnostic Test: Withdrawal of blood samples for D-Dimer — Blood samples are withdrawn at birth via cord blood and at postnatal 3rd and 7th days via umbilical catheter in order to test for D-dimer levels.
Diagnostic Test: Withdrawal of blood samples for Fibrinogen — Blood samples are withdrawn at birth via cord blood and at postnatal 3rd and 7th days via umbilical catheter in order to test for Fibrinogen levels.
Diagnostic Test: Echocardiographic Examination — At postnatal 3rd, 7th and 14th days, Ductus Arteriosus will be echocardiographically examined to obtain calculations and confirm status of ductal patency or closure.

SUMMARY:
The aim of this study is to investigate whether there is a relationship between echocardiographic measurements regarding closure of PDA and serum D-Dimer and Fibrinogen levels in premature infants born before 32nd gestational week and weighing less than 1500 grams.

DETAILED DESCRIPTION:
Ductus arteriosus (DA) is located between the main pulmonary artery and descending aorta in embryonal life, with dense spiral-located smooth muscle cells in the media layer, and the intima layer is thicker than the aorta. It must be open in fetal life; in this way, the blood flowing from the right ventricle to the collapsed lungs is directed to the descending aorta. DA usually closes "functionally" by constriction of the media during the first three days after labor. In the second week after birth; endothelial folding, subendothelial proliferation and coagulation processes results in "anatomical" permanent closure.

When not closed, patent ductus arteriosus (PDA) is formed resulting in shunting from aorta to pulmonary artery. Probability of patency is inversely related with birth weight. Risk of pulmonary edema, pulmonary hemorrhage, bronchopulmonary dysplasia and loss of pulmonary function increases due to increased pulmonary flow from left to right shunt. Renal, mesenteric and cranial blood supply are impaired due to reduced peripheral circulation. As a result, impaired renal function and necrotizing enterocolitis may develop. Risk of intracranial hemorrhage, cerebral hypoxia and premature retinopathy due to variable blood supply. It has been associated with increased mortality in newborns due to increased morbidity. On physical examination, hyperdynamic precordium, viable pulses and left ventricular hypertrophy are observed. Large PDAs are characterized by prominent pulmonary conus, increased pulmonary vascularization and cardiomegaly on telecardiography.

Diagnosis of PDA is confirmed by echocardiography. Symptomatic PDA treatment and follow-up is mostly followed by echocardiography. Detailed echocardiographic examination can only be performed by a Pediatric Cardiologist, but it is not possible to evaluate DA at any time. It is necessary to benefit from significant changes in specific hematological parameters that may accompany DA closure in order to detect and predict these conditions.

One of the main mechanisms involved in anatomic permanent closure in DA is platelet aggregation and coagulation. To the best of our knowledge, there is no study in the literature investigating whether there is a relationship between Fibrinogen and D-dimer levels and anatomical closure of DA. It is postulated that circulating fibrinogen levels will decrease and D-dimer levels increase as a by-product due to thrombosis in the lumen during DA closure. It is predicted that in infants in whom DA does not close and remain open, fibrinogen levels will be higher and D-dimer levels will be lower than infants in whom DA is closed. It is also suggested that echocardiographic DA measurements will correlate with serum Fibrinogen and D-Dimer levels.

The aim of this study is to investigate whether there is a relationship between echocardiographic measurements regarding closure of PDA and serum D-Dimer and Fibrinogen levels in premature infants born before 32nd gestational week and weighing less than 1500 grams.

ELIGIBILITY:
Inclusion Criteria:

premature newborns born before 32nd gestational week and weighing less than 1500 grams.

Exclusion Criteria:

Babies with:

* Major congenital anomalies
* Chromosomal anomalies
* Inborn errors of metabolism
* Hypoxic ischemic encephalopathy
* Disseminated intravascular coagulation
* Unstable hemodynamic status
* Severe neonatal sepsis
* Who died in time frame of postnatal 14 days
* Patients who are not volunteered to participate

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: otherwise healthy premature newborns born before 32nd gestational week and weighing less than 1500 grams.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rise in D-dimer blood levels during Ductus Arteriosus closure from postnatal day 0 to postnatal 3rd and 7th days | postnatal 0 - 14 days
  It is postulated that circulating D-dimer levels will increase gradually as a by-product due to thrombosis in the lumen during DA closure from postnatal day 0 to postnatal 3rd and 7th days. It is predicted that D-dimer levels will be lower in infants in whom DA does not close than in infants whom DA is closed. Blood samples are withdrawn accordingly at birth via cord blood and at postnatal 3rd and 7th days via umbilical catheter in order to test for D-dimer levels.
Fall in Fibrinogen blood levels during Ductus Arteriosus closure from postnatal day 0 to postnatal 3rd and 7th days | postnatal 0 - 14 days
  It is postulated that circulating fibrinogen levels will fall gradually due to thrombosis in the lumen during DA closure from postnatal day 0 to postnatal 3rd and 7th days. It is predicted that fibrinogen levels will be higher in infants in whom DA does not close than in infants whom DA is closed. Blood samples are withdrawn accordingly at birth via cord blood and at postnatal 3rd and 7th days via umbilical catheter in order to test for fibrinogen levels.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Tolga Çelik, Study Chair — Hacettepe University; Alper Aykanat, Principal Investigator — Hacettepe University; İlker Ertuğrul, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tay SP, Cheong SK, Boo NY. Circulating tissue factor, tissue factor pathway inhibitor and D-dimer in umbilical cord blood of normal term neonates and adult plasma. Blood Coagul Fibrinolysis. 2003 Feb;14(2):125-9. doi: 10.1097/00001721-200302000-00002. PMID 12632021
- [Background] Sehgal A, Paul E, Menahem S. Functional echocardiography in staging for ductal disease severity : role in predicting outcomes. Eur J Pediatr. 2013 Feb;172(2):179-84. doi: 10.1007/s00431-012-1851-0. Epub 2012 Oct 11. PMID 23052621